CLINICAL TRIAL: NCT06634628
Title: First in Human Adaptive Study to Investigate the Kinetic Properties of the Novel PET Radioligand [11C]CHDI-00491009 and Its Suitability for Quantification of Aggregated Mutant Huntingtin in the Brains of People With Huntington's Disease
Brief Title: iMagemHTT- 009- FIH Evaluation of Novel Mutant Huntingtin PET Radioligand [11C]CHDI-00491009
Acronym: iMagemHTT-009
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CS-5583
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Huntington Disease; HD; PET Tracer; Positron Emission Tomography; Radioligand; Imaging; mHTT; Huntington's; Huntington's Disease
Keywords: iMagemHTT; Huntington Disease; HD; PET Tracer; Positron Emission Tomography; radioligand; imaging; mHTT; huntingtin; Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: People with Huntington's disease (PwHD) compared to healthy controls (HC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Radioligand [11C]CHDI-00491009 3 HCs - MRI and PET Radioligand is administered 1x each person
  Interventions: Radiation: Radioligand [11C]CHDI-00491009
- Cohort 2 (Experimental): Radioligand [11C]CHDI-00491009 6 HCs - MRI and PET 6 PwHD HD-ISS Stage 2 - MRI and PET Radioligand administered 2x (TRT) for 3 HCs and 3 PwHD Radioligand administered 1x for 3 HCs and 3 PwHD In addition, optional CSF collection for all PwHD
  Interventions: Radiation: Radioligand [11C]CHDI-00491009
- Cohort 3 (Experimental): Radioligand [11C]CHDI-00491009 6 HCs - MRI and PET 6 PwHD HD-ISS Stage 3 - MRI and PET Radioligand administered 1x for 6 HCs and 6 PwHD In addition, optional CSF collection for all PwHD Depending on previous results and as decided by executive committee, TRT may be included in Cohort 3. A TRT decision would include one extra imaging session per participant (i.e., radioligand administered 2x per participant.)
  Interventions: Radiation: Radioligand [11C]CHDI-00491009

INTERVENTIONS:
Radiation: Radioligand [11C]CHDI-00491009 — Intravenous injection of radioligand in the arm with PET imaging of the brain.

SUMMARY:
This is a FIH (first-in-human) study to evaluate the clinical utility of the radioligand [11C]CHDI-00491009 as a PET tracer that binds specifically to mutant huntingtin (mHTT) aggregates in Huntington's disease (HD).

The study is divided into three cohorts defined by the Huntington's Disease Integrated Staging System (HD-ISS): Cohort 1 - initial tracer validation (3 healthy controls (HCs)); Cohort 2 - target validation and test-retest variability (6 HD-ISS Stage 3 participants and 6 age and biological sex-matched HCs); Cohort 3 - target sensitivity (6 HD-ISS Stage 2 participants and 6 age and biological sex-matched HCs). An interim analysis (IA) will be conducted after the completion of each cohort, followed by a final analysis for the study.

In addition to imaging, exploratory biomarkers, including somatic instability index, soluble mHTT and total huntingtin (HTT), will be assessed. All participants with HD (PwHD) will have an additional blood sample drawn at the screening visit to assess the somatic instability index and will also be invited to provide an optional cerebrospinal fluid (CSF) sample for measurement of soluble mHTT and total HTT.

DETAILED DESCRIPTION:
The PET radioligand [11C]CHDI-00491009 will be evaluated for its suitability for use in clinical research to quantify mHTT aggregates in PwHD. The PET radioligand is administered as a microdose of <0.5 μg and will not be administered at pharmacological doses. This study has an adaptive and modular design with three consecutive cohorts. The execution of each cohort is dependent on results from the previous cohort.

Cohort 1- Screening and imaging of 3 HCs followed by an interim analysis to evaluate the tracer kinetics without target expression (mHTT) to identify potential brain penetrating radiometabolites or other issues that may interfere with accurate quantification. If the kinetics are found to be favorable during the IA and there are no other confounding issues that may interfere with accurate quantification, then the study will proceed to target validation with Cohort 2.

Cohort 2- Screening and imaging of 6 HD-ISS Stage 3 participants and 6 age and biological sex-matched HCs. 3 HCs and 3 HD participants from Cohort 2 will be imaged twice to determine variability between scans (test-retest; TRT). An IA will be conducted after completion of Cohort 2 that will establish the optimal method for quantification of signal and endpoint, as well as evaluating the tracer binding in HD compared to HC participants and determining the TRT reproducibility. Results will then be reviewed and a go/no-go decision will be made; if [11C]CHDI-00491009 demonstrates favorable kinetic and binding properties and go criteria are met, the study will proceed to Cohort 3 evaluation. Otherwise, the study will be terminated.

Cohort 3- Screening and imaging of 6 HD-ISS Stage 2 participants and 6 age and biological sex-matched HCs. An IA will be conducted after completion of Cohort 3 to evaluate binding in HD compared to HC participants.

This adaptive study design allows for review and analysis after each cohort. The progression through each level of analysis will indicate whether [11C]CHDI-00491009 is a suitable radioligand to measure mHTT aggregate levels with sufficient sensitivity to become a potential disease progression and efficacy biomarker in Huntington's disease.

ELIGIBILITY:
Inclusion Criteria:

PwHD HD-ISS Stages 2 and 3 and HC participants who:

1. Are female or male adults, age 18-64 years old, inclusive.
2. Have body mass index (BMI) between 19 and 35, inclusive.
3. Have capacity to give full informed consent in writing and have read and signed the informed consent form (ICF).
4. Are able to comply with study procedures, including fasting and blood sampling.
5. Are able and willing to travel to the imaging center in Leuven, Belgium.
6. Are willing to comply with the use of adequate contraceptive measures.

   HD-ISS Stage 2 participants who:
7. Have a huntingtin gene CAG expansion between 40 and 50, inclusive; and
8. Are classified within HD-ISS Stage 2 per the HD-ISS criteria using HD-ISS Modified Stage calculator.
9. Have a PIN score of 0.47 to 1.84 [prognostic index normed for HD (PIN) where PIN = (PIHD - 883)/1044 where PIHD = 51 x TMS + (-34) x SDMT + 7 x Age x (CAG - 34) (TMS is the UHDRS Total Motor Score, and SDMT is the UHDRS Symbol Digit Modalities Test)].

HD-ISS Stage 2 participants who:

7. Have a huntingtin gene CAG expansion between 40 and 50, inclusive; and 8. Are classified within HD-ISS Stage 2 per the HD-ISS criteria using HD-ISS Modified Stage calculator.

9. Have a PIN score of 0.47 to 1.84 [prognostic index normed for HD (PIN) where PIN = (PIHD - 883)/1044 where PIHD = 51 x TMS + (-34) x SDMT + 7 x Age x (CAG - 34) (TMS is the UHDRS Total Motor Score, and SDMT is the UHDRS Symbol Digit Modalities Test)].

HC participants who:

13. Have no known family history of HD; or 14. Have a known family history of HD and have been tested for the huntingtin gene CAG expansion and are not at genetic risk for HD (CAG < 36).

15. Age match (+/- 5 years) and biological sex match to each HD participant in Cohort 2 and Cohort 3 (except for Cohort 1, no matching).

Exclusion Criteria:

PwHD HD-ISS Stages 2 and 3 and HC participants who:

1. Are currently participating in, or are less than 30 days after completing participation in, other therapeutic or imaging studies.
2. Have previously participated in a PET imaging study in the past 12 months that, cumulatively with the current study, will exceed annual regulatory limits for radiation exposure.
3. Have any disease, condition, or concomitant medication that significantly compromises the function of the body systems and that, in the opinion of the Investigator, might interfere with the conduct of the study or its interpretation.
4. Are pregnant and breastfeeding females.
5. Have concomitant use of antiplatelet or anticoagulant therapy (inclusive of acetylsalicylic acid).
6. Have a bleeding disorder.
7. Have a needle phobia.
8. Have any metal objects present in the body that are incompatible with MRI.
9. Have metal objects present in the body that are compatible with MRI and are located in the head or neck.
10. Have any clinically significant results on safety laboratory tests that, in the opinion of the Investigator, would either put the participant at risk or interfere with the conduct of the study or interpretation of data. These tests include, but are not limited to:

    * a. positive results for HBsAg, HepC, HIV-1 or HIV-2 (will also be reported as required by local/national regulations),
    * b. clinically significant, abnormal results for safety laboratory tests.

    PwHD participants who:
11. If they are using any antidepressant, psychoactive, psychotropic or other medications or nutraceuticals used to treat HD, the use of inappropriate (e.g., non-therapeutically high) or unstable dose within 30 days prior to participation.

    HC participants who:
12. Have a family history of HD and have not been tested for the huntingtin gene (CAG) expansion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The VT (volume of distribution total) of the PET radioligand will be measured with PET imaging. | Time Frame: Single point measure - 90 minutes scan
  The VT (volume of distribution total) of the PET radioligand will be measured with PET imaging. [Time Frame: Single point measure - 90 minutes scan] VT is derived from the data collected during each PET scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaire Ziekenhuizen Leuven/ UZ Leuven/ UZL, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided